CLINICAL TRIAL: NCT06109740
Title: Probiotics For The Prevention of Antibiotics Associated Diarrhea in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Collaborators: Amerifit Brands Inc (Industry)
Responsible Party: Principal Investigator, Allison Chung, Associate Professor, University of South Alabama
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-218
Record Dates: First submitted 2023-10-20; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Antibiotic-associated Diarrhea
Keywords: Pediatric; PICU
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Prospective randomized, double-blind, placebo-controlled crossover trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Matching placebo. Dispensed from pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus GG (Experimental): Probiotic nutritional supplement
  Interventions: Dietary Supplement: lactobacillus GG
- Placebo capsule (Placebo Comparator): Matching placebo capsule
  Interventions: Dietary Supplement: lactobacillus GG

INTERVENTIONS:
Dietary Supplement: lactobacillus GG — probiotic

SUMMARY:
The goal of this prospective trial is to learn about lactobacillus use in critically ill pediatric patients. The main question[s] it aims to answer are:

* Is lactobacillus GG effective in preventing antibiotic associated diarrhea in the PICU
* Is lactobacillus safe in critically ill pediatric patients Participants will be randomized to lactobacillus GG vs placebo while on antibiotics

If there is a comparison group: Researchers will compare lactobacillus GG to see if it prevents antibiotic associated diarrhea.

DETAILED DESCRIPTION:
The objective of this study was to assess the efficacy of lactobacillus GG (LGG) to prevent antibiotic-associated diarrhea (AAD) in the PICU.

Design:

Prospective randomized, double-blind, placebo-controlled trial

Setting:

15-20 bed PICU at University of South Alabama, Children's and Women's Hospital in Mobile, Alabama.

Patients:

Pediatric patients ≤ 17 years and required antibiotic therapy ≥ 72hrs were randomized to receive placebo or control (lactobacillus GG). Exclusion criteria included but was not limited to antibiotics ≥ 48 hours prior, prior probiotics, pre-existing diarrhea, laxative therapy, immunocompromise, and GI disorders.

Interventions:

Treatment with LGG (30 x 109 CFU) or a matching placebo capsule was administered twice daily, initiated within 24 hours of starting antibiotic therapy and continued for the duration of therapy.

Measurements:

Diarrhea was defined as stools >200 mL or 200 g per day in a patient over 10 kg and > 20 mL/kg/day or > 20 g/kg/day in a patient < 10 kg or 3 or more loose stools in 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to PICU
* Requiring > 72 hrs of antibiotic therapy
* < 17 years
* Able to administer oral LGG or placebo

Exclusion Criteria:

* Antibiotics 48 hours prior to hospital admission
* Probiotic use within 7 days of admission
* Pre-existing diarrhea at time of hospital admission or 24 hours prior to admission
* Laxative therapy at time of admission or 48 hours prior to admission
* HIV with CD4 < 250
* Established immunologic deficiencies (ANC < 100)
* Chronic steroid therapy ( > 10 days)
* GI disorders including intussusception, lower bowel disease, bowel resection, irritable bowel syndrome, ulcerative colitis, or Crohn's disease
* Status post-surgical patients with antibiotic prophylaxis (< 72 hours duration)
* NPO

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic associated diarrhea | Full time while on antibiotics and 48 hours after
  Diarrhea was defined as stools >200 mL or 200 g per day in patients over 10 kg and > 20 mL/kg/day or > 20 g/kg/day in patients < 10 kg or 3 or more loose stools in 24 hours if the stools were not able to be weighed. When patients developed diarrhea lasting more than 72 hours, they were crossed over to the alternate treatment arm.

SECONDARY OUTCOMES:
Tolerability of lactobacillus GG | 2 weeks
  Assessment of any adverse events related to lactobacillus GG

CONTACTS AND LOCATIONS:
Overall Officials: Allison Chung, Principal Investigator — University of South Alabama

IPD SHARING:
Plan to Share IPD: No
Only deidentified data